CLINICAL TRIAL: NCT05417503
Title: Acute Effects of NIV on Peripheral Muscle Function and Aerobic Performance in Patients With Chronic Obstructive Pulmonary Disease: a Piloty Study
Brief Title: Non Invasive Ventilation on Peripheral Muscle Function and Aerobic Performance
Acronym: NIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Patri-cia Angelica de Miranda Silva Nogueira, Professora associada da UFRN, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1a2b3c4d5e6f7g
Record Dates: First submitted 2022-06-03; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Skeletal muscle; Non-Invasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bi-level (Experimental)
  Interventions: Other: Non-invasive ventilation bi-level
- placebo (Placebo Comparator)
  Interventions: Other: Non-invasive ventilation placebo

INTERVENTIONS:
Other: Non-invasive ventilation bi-level — For the NIV intervention, two levels of positive airway pressure (bi-level) were used: the positive inspiratory airway pressure (IPAP) was fixed at 6 cmH2O (centimeters of water), which could be gradually increased up to 14 cmH2O (2 cmH2O every minute), depending on the patient's comfort. and gradually increased to 14 cmH2O (2 cmH2O every minute), While the expiratory airway pressure (EPAP) was set at 3 cmH2O, it could be gradually increased up to 7 cmH2O (1 cmH2O every minute), depending on the patient's comfort.while expiratory airway pressure (EPAP) was fixed at 3 cmH2O and gradually increased to 7 cmH2O (1 cmH2O every minute).
  Arms: bi-level
Other: Non-invasive ventilation placebo — The same pressure chosen by the subject during adaptation was used in the placebo intervention; however, a T tube was connected between the equipment and the circuit, creating a leak and leaving the circuit open. The tube characteristics were: 22 x 18 x 22 mm nebulizer T-connector.
  Arms: placebo

SUMMARY:
Background: Non-invasive ventilation (NIV) reduces respiratory load and demands on peripheral muscles. Methods: This study aims to evaluate the acute effects of bi-level NIV on peripheral muscle function during isokinetic exercise and aerobic performance in chronic obstructive pulmonary disease (COPD) patients. This is a pilot crossover study performed with a non-probabilistic sample of 14 moderate to very severe COPD patients. Procedures carried out in two days. Dyspnea, quality of life, lung function, respiratory muscle strength, functional capacity (6-minute walk test - 6MWT), and isokinetic assessment of the quadriceps were assessed. Blood samples (lactate, lactate dehydrogenase, and creatine kinase concentration) were also collected. Right after, NIV was performed for 30 minutes (bi-level or placebo, according to randomization) followed by new blood sample collection, 6MWT, and isokinetic dynamometer tests. Before and after evaluations, the subjective perception of dyspnea and fatigue in the lower limbs was quantified. After a wash-out period of seven days, participants returned, and all assessments were performed again.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable COPD patients (diagnosed according to the Global Initiative for Obstructive Lung Disease), of both sexes, without exacerbation or changes in medication for at least one month before the study, and no dyspnea during daily activities (grades 2, 3, and 4 of the Medical Research Council - MRC scale) were included.

Exclusion Criteria:

* Those with a diagnosis of neoplasia, orthopedic or neurological conditions affecting exercise capacity, peripheral arterial obstructive disease, heart failure, kidney or liver disease, did not adapt, or failed to complete the study procedures, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Lung function | change from baseline and 30 minutes after intervention
  Lung function was assessed using a spirometer (Koko Digidoser, Longmont, USA), according to the American Thoracic Society/European Throracic Society recommendations14. At least three tests were performed, with a variation of less than 5%, and the highest value obtained was compared with predicted values for the Brazilian population.
Respiratory muscle strength | change from baseline and 30 minutes after intervention
  Respiratory muscle strength was assessed using a digital manometer (MVD 300 - Brazil). Maximum inspiratory and expiratory pressures were performed from residual volume and total lung capacity, respectively, and values were compared with previously reference values for the Brazilian population
Functional capacity | change from baseline and 30 minutes after intervention
  The 6-minute walk test (6MWT) was performed in a flat 30-m corridor, according to the ATS recommendations17. Subjects were instructed to keep walking for six minutes, and standardized verbal incentives were given each minute. The perception of dyspnea (using the 10-point Borg scale) were assessed at rest, at the end of the 6MWT, and two minutes after the test. In this test, the walked distance (in meters) was considered for analysis.
COPD Assessement Test | change from baseline and 30 minutes after intervention
  The Portuguese version of the COPD Assessment Test (CAT) questionnaire was used to assess the quality of life. Subjects were instructed to choose only one option in each item of the questionnaire (cough, phlegm, chest tightness, breathlessness, limited activities, confidence leaving home, sleeplessness, and energy). Item scores range from 0 to 5 points resulting in a total score ranging from 0 to 40 points. The clinical impact of COPD was assessed according to the following stratification: mild (6-10), moderate (11-20), severe (21-30), and very severe (31-40)20.
Disease severity | change from baseline and 30 minutes after intervention
  COPD severity was assessed using the BODE index (body mass index [B], degree of airway obstruction [O], dyspnea [D], and exercise capacity [E]). For each variable, the following scores were assigned: body mass index (BMI), from 0 to 1 point; degree of airflow obstruction (FEV1% predicted), from 0 to 3 points; dyspnea (MRC scale), from 0 to 3 points; exercise capacity (walked distance in the 6MWT), from 0 to 3 points. The final score of the index ranges from 0 to 10, with higher scores indicating greater disease severity.

SECONDARY OUTCOMES:
Quadriceps femoris performance | change from baseline and 30 minutes after intervention
  QF (Quadriceps femoris) strength was evaluated with subjects performing 20 repetitions at the same speed. The protocol established was designed to reach a fatigue threshold in the QF muscle. Dyspnea and perceived level of exertion (Borg scale) were also assessed before and after isokinetic evaluation.
Biochemical analyzes | change from baseline and 30 minutes intervention
  Before and after procedures, venous blood samples were collected by a blinded experienced pharmacist to analyze lactate, LDH enzyme, and CK (creatine kinase) concentration. Samples were processed, centrifuged at 3000 rpm for 15 minutes at room temperature. The serum concentration was assessed using a specific enzyme kit for each biomarker, following manufacturer's recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Nogueira, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No